CLINICAL TRIAL: NCT01498458
Title: Phase I Study to Assess the Optimal Dose for Pazopanib in Combination With Capecitabine in Patients With HER2-negative, Metastatic Breast Cancer (PazoX)
Brief Title: Pazopanib in Combination With Capecitabine in Patients With Metastatic Breast Cancer
Acronym: PazoX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBG 62; 2010-019510-25 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2014-09

CONDITIONS: Metastatic Breast Cancer
Keywords: German Breast Group; GBG Forschungs GmbH; GBG; GBG 62; PazoX; Breast Cancer; Metastatic Breast Cancer; Pazopanib; Abraxane; Capecitabine; Xeloda
MeSH Terms: conditions — Breast Neoplasms | interventions — pazopanib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pazopanib plus capecitabine (Experimental)
  Interventions: Drug: Pazopanib plus capecitabine

INTERVENTIONS:
Drug: Pazopanib plus capecitabine — Patients will receive pazopanib tablets once daily at a dose according to the allocated dose level:
  * dose level I: 400 mg
  * dose level II: 600 mg
  * dose level III: 800 mg
  In addition patients receive capecitabine at the same oral dose for all dose levels with 1600 mg/m2 on days 1 to 14 every 3 weeks.
  Treatment will be given until disease progression or unacceptable toxicity of the study drug, or withdrawal of consent of the patient.
  Six patients will be recruited in each dose level. If less than 2 out of 6 patients experience a DLT within the first 2 cycles (weeks 1 to 6), the next dose level is started. Once the MTD is established, additional 6 patients will be included into this dose level to further characterise the safety of the dose regimen.
  If it is reported, that two patients had a DLT, all patients are informed about it and the dose level immediately reduced by one dose level.

SUMMARY:
Angiogenesis is essential for the growth of large tumor. A number of anti-angiogenic agents are currently under development. Bevacizumab, a humanised monoclonal antibody to vascular endothelial growth factor (VEGF), has been shown to improve disease free survival in first line metastatic breast cancer when associated with chemotherapy 1. Results of a randomised phase II trial combining sorafenib, a tyrosine kinase inhibitor targeting multiple tyrosine kinases including VEGFR1, VEGFR2, VEGFR3, with capecitabine have recently been reported 2. Compared to capecitabine plus placebo, progression-free survival in the capecitabine + sorafenib arm was significantly increased from 4.1 months to 6.4 months. Toxicities were also increased, with an incidence rate of grade 3/4 hand foot syndrome of 45% in the capecitabine + sorafenib arm compared to 13% in the capecitabine + placebo arm. The increased toxicity will most likely limit the clinical use of this regimen.

Pazopanib is a potent, multi-targeted TKI of VEGFR-1, -2, -3, PDGFR-α and -β and c-kit and has recently been approved for the treatment of renal cell cancer in the U.S. In the EU, a positive opinion has been issued by the European Medicines Agency.

A phase II study of GW786034 (pazopanib) in patients with recurrent or metastatic invasive breast carcinoma included 19 patients after a maximum of 2 lines of chemotherapy for advanced disease 3. Pazopanib 800 mg daily was given continuously.

A clinically significant rate of stable disease (58%) was detected with a median TTP of 5.3 months (95% CI: 1.8 - 9.0 months). Four patients treated with pazopanib had SD for ≥ 6 months, for a clinical benefit rate (CBR), defined as rate of SD for ≥ 6 months or CR or PR, of 5/19 (26%), which is at least comparable to sunitinib and bevacizumab (CBR 16% and 17%, respectively).

The pivotal study of full dose (800 mg) daily pazopanib in renal cell cancer reported hand foot syndrome of all grades in only 6% of patients 4. The optimally tolerated regimen (OTR) of pazopanib was determined when administered in combination with capecitabine and oxaliplatin in patients with advanced CRC 5. In patients who received capecitabine (850 mg twice daily) plus 800 mg once daily pazopanib combined with oxaliplatin, the incidence of hand foot syndrome of all grades was 24%.

The present study will investigate the combination of pazopanib and capecitabine in advanced or metastatic breast cancer with the aim to develop a new treatment option with increased efficacy and tolerability.

DETAILED DESCRIPTION:
Primary Objective:

To assess the maximum tolerated dose (MTD) of pazopanib in combination with capecitabine as treatment for metastatic HER2-negative breast cancer.

Secondary Objective:

1. To determine the dose-limiting toxicity (DLT).
2. To determine the compliance and toxicity of the combination.
3. To determine the objective response rate (ORR) and clinical benefit rate (CBR) in patients with measurable disease.
4. To determine the duration of response.
5. To determine the progression-free survival (PFS).
6. To determine the predictive value for response of serum markers such as VEGF.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
* Complete baseline documentation must be submitted via the web-based data collection system MedCODES to the GBG Forschungs GmbH.
* Diagnosis of advanced or metastatic HER2-negative breast cancer. HER2-negative is defined as HercepTest IHC 0-2+ or FISH negative (ratio < 2.2).
* At least one prior endocrine or one non-capecitabine-containing chemotherapy treatment for metastatic/advanced disease.
* Documented progression of either a measurable, or a non-measurable lesion according to the RECIST criteria, or a new lesion.
* Complete radiological and clinical tumor assessment within 4 weeks prior to registration performed as clinically indicated.
* Age => 18 years.
* Karnofsky Performance Status index => 60%.
* Laboratory requirements: Absolute neutrophil count (ANC) => 1.5 x 109/L, Platelets => 100 x 109/L, Hemoglobin => 9 g/dL (=> 5.6 mmol/L), Prothrombin time (PT) or international normalised ratio (INR) =< 1.2x UNL (upper normal limit), Partial thromboplastin time (PTT) =< 1.2x UNL, Total bilirubin < 1.5x UNL, ASAT (SGOT) and ALAT (SGPT) =< 2.5x UNL (concomitant elevations in serum bilirubin and ASAT/ALAT above 1.0x UNL are not permitted), The calculated creatinine clearance should be => 50 mL/min), Urine Protein to Creatinine Ratio (UPC) < 1 (if UPC => 1, then 24-hour urine protein must be < 1 g).
* Normal cardiac function confirmed by ECG; corrected QT interval (QTc) < 480 msec using Bazett's formula.
* A female either of:Non-childbearing potential i.e., physiologically incapable of becoming pregnant because of history of hysterectomy, bilateral oophorectomy (ovariectomy), bilateral tubal ligation or postmenopausal status.

Childbearing potential with a negative serum pregnancy test within 2 weeks prior to registration, preferably as close to the first dose as possible, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow: An intrauterine device with a documented failure rate of less than 1% per year, Vasectomised partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female, Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product, Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

* Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

* Known or suspected hypersensitivity reaction to the investigational compounds or incorporated substances.
* Last metastatic treatment with capecitabine, 5-FU, bevacizumab, sunitinib, sorafenib, or other antibodies or tyrosine kinase inhibitors with anti-angiogenic activity. Investigational therapies within 14 days or five half-lives of the drug (whichever is longer) prior to first dose of pazopanib.
* Any ongoing toxicity from prior anti-cancer therapy that is grade >1 and/or that is progressing in severity, except alopecia.
* Surgery or tumor embolisation within 28 days prior to the first dose of pazopanib. At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiated field or there must be pathological proof of progressive disease.
* Concurrent immuno-biological or hormonal therapy for cancer.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug.
* Life expectancy less than 3 months.
* History of thyroid autoimmune disease or thyroid disorders with thyroid values out of standard range
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to: Active peptic ulcer disease, Known intraluminal metastatic lesion/s with risk of bleeding, Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation, History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* Severe liver dysfunction
* Grade 3 or 4 diarrhea.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: Malabsorption syndrome, Major resection of the stomach or small bowel.
* Presence of uncontrolled infection.
* History of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting, Myocardial infarction, Unstable angina, Coronary artery bypass graft surgery, Symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA), Poorly controlled hypertension (defined as systolic blood pressure [SBP] of ≥ 160 mmHg or diastolic blood pressure [DBP] of ≥ 90 mmHg).

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.

BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP/DBP values from each BP assessment must be < 160/95 mmHg in order for a subject to be eligible for the study (see Section 9.6.1 for details on BP control and re-assessment prior to study enrollment).

* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
* Evidence of active bleeding or bleeding diathesis including, but not limited to: Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major), Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels, Hemoptysis prior to 6 weeks of first dose of study drug, Blood transfusion within 7 days of study entry.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GBG Forschungs GmbH, Neu-Isenburg, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 patients were registered in the study but patient number 9 withdrew consent immediately without receiving any Pazopanib.
Groups:
- Pazopanib Plus Capecitabine: The baseline refers only to the 8 patients who received Pazopanib.
Period: Overall Study
Arm/Group | Pazopanib Plus Capecitabine
Started | 8 (9 patients took part in the study of which 8 received pazopanib.)
Completed | 1 (only 1 patient was in the study at the end. 7 left due to Adverse Events or Investigators Decision.)
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Pazopanib Plus Capecitabine: pazopanib plus capecitabine
Arm/Group | Pazopanib Plus Capecitabine
Number analyzed (Participants) | 8
Age, Customized [Number; unit: participants]
  premenopausal | 1
  Postmenopausal | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
ECOG [Number; unit: participants] — ECOG Status refers to the Eastern Cooperative Oncology Group scale . These scales and criteria are used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis...Grade 0 Fully active
  * Grade 1 restricted in physically strenuous activity
  * Grade 2 Ambulatory and capable of all selfcare
  * Grade 3 Capable of only limited selfcare
  * Grade 4 Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  * Grade 5 Dead
  participants
    ECOG 0 | 6
    ECOG 1 | 2
T status [Number; unit: participants] — T status describes the size of the original (primary) tumor and whether it has invaded nearby tissue,,,T1 - The tumour is 2 centimetres (cm) across or less...T2 - The tumour is more than 2 centimetres, but no more than 5 centimetres across...T3 - The tumour is bigger than 5 centimetres across...T4 refers to inflamatory breast cancer....Tis means DCIS(ductal carcinoma in situ...The tumors are all breast cancer tumors as the study has to do with breast cancer.
  participants
    T1 | 2
    T2 | 3
    T3 | 0
    T4 | 2
    Tis | 1
N Status [Number; unit: participants] — N status is a categorisation of the number of lymph nodes..N0 - No cancer cells found in any nearby nodes...N1 is when 1 to 3 lymph nodes are found.....N2 is when 4 to 9 lymph nodes are found....N2 is when greater than 9 lymph nodes are found
  participants
    N0 | 2
    N1 | 5
    N2 | 0
    N3 | 1
Grading [Number; unit: participants] — Grading is a measure of the cell appearance in tumors and other neoplasms in pathology...Grade 1 Well differentiated (Low grade)...
  Grade 2 Moderately differentiated (Intermediate grade)... Grade 3 poorly differentiated (High grade)
  participants
    G1 | 0
    G2 | 5
    G3 | 3
Hormone Receptor Status [Number; unit: participants]
  ERneg/PRneg | 2
  ERneg/PRpos | 1
  ERpos/PRneg | 2
  ERpos/PRpos | 3
HER2 Status [Number; unit: participants]
  Her2 Negative | 8
  Her2 Positive | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerable Dose (MTD) of Pazopanib
Description: The maximum tolerated dose (MTD) is defined as the highest dose level with DLT in no more than 1 out of 6 patients. A maximal tolerated dose (MTD) could not be established.
Time Frame: 3 years
Measure: Number; unit: mg
Groups:
- Pazopanib Plus Capecitabine: A maximal tolerated dose (MTD) could not be established. The study was stopped after 8 patients.
Arm/Group | Pazopanib Plus Capecitabine
Number analyzed (Participants) | 8
mg | NA — no patients reached the second dose level.

2. Secondary Outcome: Dose-limiting Toxicity (DLT)
Time Frame: 3 years
Measure: Number; unit: participants
Groups:
- Pazopanib Plus Capecitabine: The following DLTs resulted in permanent discontinuation of the study therapy: hypertension, (DLT 1), mucositis CTC grade 3, hand-foot-syndrome CTC grade 3, increase of liver enzymes (GOT,- and GPT) CTC grade 2 (DLT 2), and increase of liver enzymes (GOT-, GPT) CTC grade 3 (DLT 3).
Arm/Group | Pazopanib Plus Capecitabine
Number analyzed (Participants) | 8
participants | 5

3. Secondary Outcome: Hematological Toxicity of the Combination of Pazopanib and Capecitabine
Time Frame: 3 years
Measure: Number; unit: Number of cycles
Groups:
- Pazopanib + Capecitabine: Pazopanib and Capecitabine
Arm/Group | Pazopanib + Capecitabine
Number analyzed (Participants) | 8
Number of cycles
  Anemia Grade 1 to 4 | 88
  Leucopenia Grade 1 to 4 | 55
  Number of Cycles | 132

4. Secondary Outcome: Other Toxicity of the Combination of Pazopanib and Capecitabine
Time Frame: 3 years
Population: 6 patients experience 6 Serious Adverse Reactions
Measure: Number; unit: participants
Groups:
- Pazopanib Plus Capecitabine: pazopanib together with capecitabine
Arm/Group | Pazopanib Plus Capecitabine
Number analyzed (Participants) | 8
participants
  Hepatotoxicity | 3
  Hypertension | 1
  Pancreatectomy | 1
  Thrombocytopenia | 1

5. Secondary Outcome: Objective Response Rate (ORR)
Description: To determine the objective response rate (ORR) in patients with measurable disease. ORR consists of complete response and partial response according to the RECIST criteria. Complete Response refers to the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to less than 10 mm. Partial Response refers to an at least 30 percent decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 3 years
Population: All patients are included when determining this rate.
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib Plus Capecitabine
Number analyzed (Participants) | 8
percentage of participants | 0

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: To determine the clinical benefit rate (CBR) in patients with measurable disease. CBR consists of complete response , partial response, and stable disease lasting greater than 24 weeks. All patients are included when determining this rate. 2 patients were on study treatment for a long time.Hence the outcome rate of 25 percent ( 2 from 8 patients)
Time Frame: 3 years
Population: All patients are included when determining this rate.
Measure: Number; unit: percentage of participants
Groups:
- Pazopanib Plus Capecitabine: 2 patients were on study treatment for a long time.
Arm/Group | Pazopanib Plus Capecitabine
Number analyzed (Participants) | 8
percentage of participants | 25

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Pazopanib Plus Capecitabine: There was only one arm in this study as this was a dose escalation study.
Arm/Group | Pazopanib Plus Capecitabine
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib Plus Capecitabine (N=8)
Hepatotoxicity (Hepatobiliary disorders) | 3
Hypertension (Cardiac disorders) | 1
Pancreatectomy (Hepatobiliary disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib Plus Capecitabine (N=8)
Fatigue (General disorders) | 8
anemia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 7
alkaline Phosphatase (Hepatobiliary disorders) | 2
ASAT (Hepatobiliary disorders) | 7
Bilirubinaemia (Hepatobiliary disorders) | 3
Fatigue CTC grade 3 (General disorders) | 1 (1)
Nausea CTC grade 3 (Gastrointestinal disorders) | 1 (1)
Mucositis CTC grade 3 (Gastrointestinal disorders) | 1 (1)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No